CLINICAL TRIAL: NCT06839287
Title: The Effect of Relationship Psychotherapy-Based Counselling Applied to Individuals Receiving Hemodialysis Adjusment to Illness and Depression Levels: A Randomised Controlled Study
Brief Title: Interpersonal Psychotherapy-Based Counseling for Hemodialysis Patients: Effect on Adjustment and Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, TUGCE UCGUN, Research Assistant, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: BU-KA24/91-TU
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-02

CONDITIONS: Hemodialysis; Interpersonal Psychotherapy
Keywords: hemodialysis patients; depression; adjusment to illness; interpersonal psychotherapy; counseling; nursing
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: In this study, there are two groups. One of them is interventional group which participants receiving IPT for 8 weeks
Who Masked: Participant, Outcomes Assessor
Masking Description: In this study, participants will be randomly assigned to intervention and control groups. As a blinding method, it will be arranged so that the participants and the people responsible for data analysis who will make the evaluations will not know which group the participants are in (single-blind or double-blind design). Participants may know their groups due to the intervention content, but evaluations will be made with objective scales so as not to affect the study results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IPT Group (Experimental): Interpersonal psychotherapy-based counseling will be applied to indivuduals with receiving hemodialysis for 8 weeks
  Interventions: Other: Interpersonal psychotherapy-based counseling
- Control Group (No Intervention): Participants in this group will receive routine care

INTERVENTIONS:
Other: Interpersonal psychotherapy-based counseling — The first data from the individuals in the experimental and control groups will be collected after the first interview. Data will be collected from the individuals to whom interpersonal relationship therapy techniques are applied after the 8th session by face-to-face interviews. In addition, if the individuals in the experimental group have questions about psychotherapy, they will be answered. The control group will be verbally informed with the data collection form and chronic disease adaptation and depression scales and will continue to receive routine care. Data will be collected by face-to-face interviews with the control group after the first interview and 8 weeks later when they come to the dialysis center. Follow-up data of the participants will be collected again at the 3rd month after the last interview.
  Arms: IPT Group

SUMMARY:
The aim of this clinical study is to examine the effect of interpersonal psychotherapy-based counseling on adjustment to illness and depression levels in individuals receiving hemodialysis treatment.

The main questions this study aims to answer are:

Does interpersonal psychotherapy-based counseling improve the adjustment to illness in individuals receiving hemodialysis treatment? Does interpersonal psychotherapy-based counseling reduce depressive symptoms in individuals receiving hemodialysis treatment? The researchers will compare interpersonal psychotherapy-based counseling with routine care to determine its effectiveness in individuals undergoing hemodialysis treatment.

Participants:

For eight weeks, participants will receive either routine care or interpersonal psychotherapy-based counseling.

DETAILED DESCRIPTION:
INTRODUCTION AND GENERAL INFORMATION Today, increasing life expectancy increases the incidence of chronic diseases. Chronic kidney disease (CKD) is an important health problem that affects all age groups, especially young adults, burdens individuals, their families, and society, has a high risk of developing complications, leads to psychosocial problems, and has increased incidence in recent years both in the world and in our country.

The treatment of CKD varies according to the stage of the disease and the presence of chronic diseases in the individual. In treatment, high blood pressure is generally treated, renal function is protected against angiotensin-converting enzyme inhibitor drugs, plasma glucose levels are controlled in patients with diabetes, high cholesterol levels are reduced with diet and drug therapy, treatment is applied for anemia, treatment is planned for mineral and bone diseases, exercise is recommended, weight control is ensured, and the individual is encouraged to quit smoking. Renal replacement therapies (RRT) are generally applied in individuals with end-stage renal failure (ESRF). Although RRTs prolong life, they may also cause morbidity and mortality. RRT has three types: hemodialysis, peritoneal dialysis, and renal transplantation. In hemodialysis treatment, individuals diagnosed with ESRF may encounter negative effects such as being dependent on treatment programs and devices that last an average of 4-6 hours on certain days of the week (2 or 3), experiencing fear and anxiety due to machine alarms, and loss of time and workforce.

Chronic diseases are diseases that progress rapidly, negatively affect individuals' fulfillment of daily activities, have an uncertain prognosis, may lead to morbidity, affect the individual physically and psychosocially, cause economic problems, and require special care and control for a long time. CKD is one of the serious health problems included in chronic diseases. Despite the treatment methods used in the treatment of CKD, CKD causes physical and emotional problems in individuals, negatively affects their quality of life, and leads to death. Therefore, the adaptation of individuals with this disease to the disease and treatment is very important. Living with a disease such as CKD is a complex, cyclic, dynamic, and ever-changing multidimensional process in which acceptance, coping, and adaptation to the disease are necessary.

Individuals with CKD, especially individuals with ESRF, struggle with many problems in their lives, and their quality of life is negatively affected. One of the most important problems experienced by these individuals is psychosocial adaptation to the disease and complications caused by the disease. Especially hemodialysis treatment is a treatment method that causes changes in the lives of individuals. This treatment method is a process that negatively affects both individuals and families and requires new arrangements in their lives. Change in role performance, loss of health, decreased productivity, loss of power, sexual dysfunction, economic losses, limitation of independence, deterioration in body image, obligation to follow a diet, hopelessness, uncertainty about the future, disruption of family order, fear of death and loss of body functions are among the psychosocial problems experienced by these individuals.

After the acute period, adjustment difficulties and major depression are the most common mental problems in individuals with CKD. Worries about losing their health, physical strength, sexual function, independence, and productivity and experiencing a loss are effective in the occurrence of depressive symptoms in individuals with a diagnosis of CKD. There is a relationship between the deterioration of individuals' physical health and the severity of depressive symptoms. Especially individuals with insufficient psychosocial support resources have a higher risk of depressive symptoms. Depressive symptoms are a common mental problem in hemodialysis patients and are a response to the losses experienced by individuals. The physical health of individuals with a diagnosis of CKD deteriorates because of noncompliance with their diet and treatment and is thought to cause depressive symptoms. Early identification and treatment of individuals with depressive symptoms is very important in terms of continuity of hemodialysis treatment and prevention of suicides. Pharmacologic and nonpharmacologic interventions can be applied to individuals who have depressive symptoms or are diagnosed with depression during hemodialysis treatment. While antidepressants are preferred pharmacologically, nonpharmacological interventions include cognitive behavioral therapy, motivational interviewing, relaxation exercises, regular exercise, social support groups, tele-nursing programs, music therapy, light therapy, healthy nutrition, self-management, problem-solving skills and laughter therapy. When literature is examined, the use of Interpersonal Psychotherapy (IPT) in the treatment of depression seen in individuals with physical illness is increasing.

Interpersonal Psychotherapy (IPT) is a type of psychotherapy that focuses on short-term, especially interpersonal problems, and aims to reduce depressive symptoms resulting from interpersonal relationship problems and to improve interpersonal functioning. The therapy process aims to help the individual improve his/her interpersonal relationships or to change his/her expectations about these relationships. It also aims to help individuals increase their social support systems to facilitate coping with stress. The focal points of IPT are interpersonal conflicts, role changes, lack of interpersonal skills (such as social isolation), grief, and loss. There are four main aims of IPT: to facilitate the individual's grief process by listening, to help the individual complete the loss healthily, to allow the individual to express his/her experiences to others, and to support and strengthen the individual to establish new relationships. Generally applied for a short period (12-20 sessions), IPT has four basic stages. Each stage is conducted one-on-one with the individual. The aim is for the individual to recognize interpersonal relationship problems, define the problems correctly, and develop solution strategies. Although IPT was first used in the treatment of depression, it has been used in different age groups such as perinatal depression, geriatric population, and adolescents, and the treatment of different diagnoses such as dysthymia, eating disorder, bipolar disorder, posttraumatic stress disorder and anxiety disorders. Individuals with physical illness may experience loss and grief due to the disease process and the physical differences they experience and may require role change/having a new role. The IPT applied to individuals with physical illness provides benefits in coping with relationship problems arising from the experience of the illness, organizing their communication with their social environment, and having realistic expectations about their interpersonal relationships. When the literature was examined, no study was found on the use of IPT in individuals diagnosed with CKD receiving hemodialysis treatment, but there are studies examining the effectiveness of IPT in the treatment of depression accompanying physical diseases such as HIV, breast cancer, coronary artery disease, pain, chronic pain and infertility.

Today, the number of studies examining the mental problems and quality of life of hemodialysis patients is increasing. When these studies are examined, it is seen that psychoeducation, motivational interviewing, and cognitive behavioral therapy techniques are more commonly used as interventions. When literature is taken into consideration, there is no study in which IPT techniques were applied to individuals with chronic kidney disease. This study aims to determine the effect of interpersonal psychotherapy-based counseling applied to individuals receiving hemodialysis treatment on disease adaptation and depression.

Research Hypothesis:

H0-1: There is no difference between the intervention group and the control group who received interpersonal therapy-based counseling in terms of the level of adjustment to the disease in individuals receiving hemodialysis treatment.

H0-2: There is no difference in the level of depression between the intervention group and the control group who received interpersonal therapy-based counseling in individuals receiving hemodialysis treatment.

METHODS Study Design This research is designed as a randomized controlled trial (RCT) with repeated measures, including baseline (pre-test), post-test, and follow-up assessments. Participants will be randomly assigned to either the intervention group (receiving IPT-BC) or the control group (receiving standard care).

Participants The study will consist of individuals receiving hemodialysis treatment due to chronic kidney disease. The sample of the study will consist of those who received hemodialysis treatment at Başkent University Ankara Hospital Ümitköy Dialysis Center between March 2025 and July 2025 and who want to participate in the study.

Inclusion criteria:

* 18 years of age or older,
* Hemodialysis treatment for at least 6 months,
* Having no problem communicating in Turkish,
* No hearing problems and cognitive impairment,
* Openness to cooperation,
* Not diagnosed with major depression according to DSM-V and ICD-11,
* Not having an additional mental disorder,
* Not receiving any therapy or treatment,
* Receiving hemodialysis treatment at the center 3 days a week,
* Take care of yourself,
* Scoring 10 and above on the Beck Depression Inventory (scores of 10 and above indicate that the participant has depressive symptoms)
* Patients who voluntarily agree to participate in the study will be included.

Exclusion criteria:

* Changing cities during research,
* Don't want to leave the research,
* Receiving a psychiatric diagnosis during research,
* Starting therapy or treatment during the research,
* Hospitalization during research,
* Failure to attend the treatment for 2 consecutive sessions, Başkent University Statistical Consultancy and Research Center stated that at least 44 patients should be included in the study, 22 in the group receiving counseling based on interpersonal relations psychotherapy and 22 in the control group, with an effect size of f=0.25, 80% test power, 95% confidence level, and approximately equal distribution in the groups.

Research Material:

Especially with the diagnosis of physical illness, individuals think that they cannot adapt to this process and that they have a new role. Individuals with insecure attachment styles may think that there is nothing they can do after the disease diagnosis. While these individuals are working on role change, their emotions should be addressed, they should be asked to introduce their social environment, and their attachment styles should be taken into consideration. In individuals with insecure attachment styles, small role changes can cause a major crisis. The "Life Events Inventory", one of the tools of IPT, can be used to study role changes during crisis periods. In addition, it is planned to use life events inventory, interpersonal relations inventory/relationship circle techniques as well as techniques such as asking questions, explaining, informing, and receiving feedback from effective communication skills during interviews.

Intervention

IPT-BC will be delivered in eight weekly sessions, each lasting approximately 60 minutes, by a trained therapist. Sessions will be structured around four IPT phases:

1. Assessment/Initial Phase: Identification of interpersonal problems (role transitions, social isolation, grief/loss, or interpersonal disputes) using tools such as the Interpersonal Inventory and Relationship Circle. A treatment plan will be established.
2. Middle Phase: Implementation of targeted interventions based on identified interpersonal problem areas. Weekly reassessment of interpersonal dynamics.
3. Termination of acute treatment: Consolidation of treatment gains, development of coping strategies, and relapse prevention.
4. Maintenance Phase: Optional follow-up support based on individual needs, delivered through scheduled or as-needed sessions.

Control Group: Receives routine dialysis care without IPT-BC intervention.

Variables of the Study:

Independent variables: Patients' sociodemographic, disease and treatment process information (age, weight, height, marital status, educational status, occupation, income level, whether they have children, number of children, disease duration, hemodialysis treatment duration, biochemistry blood tests (potassium, phosphorus, creatinine, etc.), Kt/V ratio (for dialysis adequacy)) Dependent Variables: Scale scores (Adaptation to Chronic Diseases Scale and Beck Depression Scale scores)

Data Collection Tools:

Within the scope of the study, the Sociodemographic Data Collection Form, Adaptation to Chronic Diseases Scale, and Beck Depression Scale prepared in line with the literature on the subject will be collected.

The Process of Developing the Content of Interpersonal Psychotherapy-Based Counseling Preliminary Implementation of the Study Pre-application will be made in 10% of the sample. Necessary arrangements will be made in line with the suggestions.

Implementation Process of the Research The data of the study will be collected by the researcher through face-to-face interviews with individuals receiving hemodialysis treatment for chronic kidney disease who apply to Başkent University Ankara Hospital Ümitköy Dialysis Center and Çiğdem Dialysis Center.

In the study, the researcher will inform the patients who meet the sampling criteria about the study and those who agree to participate in the study will be randomized into experimental and control groups. A simple randomization method will be used in randomization and experimental groups and control groups will be determined using Random Allocation Software.

The first interview will be conducted with the individuals in the experimental and control groups during hemodialysis treatment in a calm and quiet environment, in a period deemed appropriate by the individual, ensuring privacy. In the first interview, which is expected to last an average of thirty minutes, the purpose of the study will be explained to the individuals. Data will be collected from the individuals in the experimental and control groups with sociodemographic information form, chronic disease adaptation scale, and Beck depression inventory, and the individuals in the experimental group will be counseled based on interpersonal relations psychotherapy.

The first data from the individuals in the experimental and control groups will be collected after the first interview. Data will be collected from the individuals to whom interpersonal relationship therapy techniques are applied after the 8th session through face-to-face interviews. In addition, if the individuals in the experimental group have questions about psychotherapy, they will be answered. The control group will be verbally informed with the data collection form and chronic disease adaptation and depression scales and will continue to receive routine care. Data will be collected by face-to-face interviews with the control group after the first interview and 8 weeks later when they come to the dialysis center. Follow-up data from the participants will be collected again in the 3rd month after the last interview.

Statistical Evaluation of Data In the study, frequency (n) and percentage (%) values will be used as descriptive statistics in the evaluation of categorical variables. Shapiro-Wilk test will be used for the conformity of numerical variables to normal distribution and as descriptive statistics; mean ± standard deviation values will be given for variables suitable for normal distribution and median (minimum-maximum) values will be given for those that do not fit the normal distribution. The appropriate hypothesis testing method planned to be used in the study was determined as a "Two-Way Analysis of Variance with Repetitions on a Single Factor" when parametric test assumptions are met. In examining whether there is a difference between groups in terms of numerical measurements, it will be examined by "Analysis of Variance" if parametric test assumptions are met, and by "Kruskal-Wallis Test" not; In examining the repetitions of numerical measurements at 3 different times, it will be examined by "Repeated measures ANOVA" if test assumptions are met, and by "Friedman test" not. In examining the relationships between variables, if the test assumptions are met, "Pearson correlation analysis" will be performed, if not, "Spearman correlation analysis" will be performed. In examining the relationship between categorical variables, "The Pearson Chi-Square Test" will be used when the test assumptions are met, and "The Fisher Exact Test" will be used when the test assumptions are not met. In all hypothesis tests, Type I error probability will be taken as α=0.05, and the SPSS v25.0 package program will be used for statistical evaluations.

Ethical Considerations Ethical approval will be obtained from the Başkent University Ethics Committee. Written informed consent will be secured from all participants. The study complies with Helsinki Declaration principles.

Expected Contributions This study will provide novel insights into the applicability of IPT-BC in CKD/HD populations, offering an alternative evidence-based psychological intervention for improving disease adaptation and mental health. If effective, IPT-BC could be integrated into standard psychosocial care for HD patients, enhancing their quality of life and treatment adherence.

ELIGIBILITY:
Inclusion Criteria:

* • 18 years of age or older,

  * Hemodialysis treatment for at least 6 months,
  * Having no problem communicating in Turkish,
  * No hearing problems and cognitive impairment,
  * Openness to cooperation,
  * Not diagnosed with major depression according to DSM-V and ICD-11,
  * Not having an additional mental disorder,
  * Not receiving any therapy or treatment,
  * Receiving hemodialysis treatment at the center 3 days a week,
  * Do not take care of yourself,
  * Scoring 10 and above on the Beck Depression Inventory (scores of 10 and above indicate that the participant has depressive symptoms)
  * Patients who voluntarily agree to participate in the study will be included.

Exclusion Criteria:

* - Having a neurological or psychiatric illness that may interfere with reading and understanding the data collection tools,
* Have received or are receiving any therapy or treatment,
* A score of 10 or less on the Beck Depression Inventory,
* Having problems in speaking/understanding Turkish,
* Changing cities during research,
* Don't want to leave the research,
* Receiving a psychiatric diagnosis during research,
* Starting therapy or treatment during the research,
* Hospitalization during research,
* Failure to attend the treatment for 2 consecutive sessions,

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-09-05 (Actual)

PRIMARY OUTCOMES:
Adaptation to Chronic Diseases Scale | five mounths
  The Adaptation to Chronic Diseases Scale was developed by Atik and Karatepe (2016) to assess the level of adaptation to the disease of individuals diagnosed with chronic diseases (heart, lung and kidney diseases, diabetes, etc.). In the scale, situations including beliefs, attitudes and behaviors experienced by individuals diagnosed with chronic diseases during the disease are specified. The scale consists of 5-point Likert type and 25 items (56). The scale has 3 sub-dimensions as Physical, Social and Psychological Adjustment. Physical Adjustment sub-dimension consists of 1st, 9th, 10th, 13th, 16th, 18th, 22-24th items, Social Adjustment sub-dimension consists of 2nd, 3rd, 5th, 7th, 17th, 19th and 25th items, Psychological Adjustment sub-dimension consists of 4th, 6th, 8th, 11th, 12th, 20th and 21st items. A maximum score of 55 and a minimum score of 11 can be obtained from the Physical Adjustment sub-dimension, a maximum score of 35 and a minimum score of 7 from the Social Adjustment

SECONDARY OUTCOMES:
Beck Depression Scale | five mounths
  The Turkish validity and reliability study of the scale developed by Beck et al. (1961) was conducted by Hisli (1989). The scale has 11 sub-dimensions measuring cognitive, 2 emotional, 2 overt behaviors, 1 interpersonal problems and 5 somatic symptoms. The scale is four-point Likert-type and consists of 21 questions in total. Each item in the scale is scored between "0-3". The lowest score is 0 and the highest score is 63. An increase in the total score obtained from the scale indicates an increase in the level of depression. Scores between 11 and 17 indicate mild depression, scores between 18 and 29 indicate moderate depression, and scores between 30 and 63 indicate severe depression (57,58). In the original format of the scale, Cronbach's alpha coefficient was found to be 0.80, and in the Turkish validity and reliability study, Cronbach's alpha value was found to be 0.74 (58).

CONTACTS AND LOCATIONS:
Locations (1):
- Başkent University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stuart S, Schultz J, Molina AP, Siber-Sanderowitz S. Interpersonal Psychotherapy: A Review of Theory, History, and Evidence of Efficacy. Psychodyn Psychiatry. 2024 Sep;52(3):370-407. doi: 10.1521/pdps.2024.52.3.370. PMID 39254940
- [Background] Summers KM, Martin KE, Watson K. Impact and clinical management of depression in patients with coronary artery disease. Pharmacotherapy. 2010 Mar;30(3):304-22. doi: 10.1592/phco.30.3.304. PMID 20180613
- [Background] Xu H, Koszycki D. Interpersonal Psychotherapy for Late-life Depression and its Potential Application in China. Neuropsychiatr Dis Treat. 2020 Aug 7;16:1919-1928. doi: 10.2147/NDT.S248027. eCollection 2020. PMID 32821108
- [Background] Karam AM, Fitzsimmons-Craft EE, Tanofsky-Kraff M, Wilfley DE. Interpersonal Psychotherapy and the Treatment of Eating Disorders. Psychiatr Clin North Am. 2019 Jun;42(2):205-218. doi: 10.1016/j.psc.2019.01.003. PMID 31046923
- [Background] Cuijpers P, Donker T, Weissman MM, Ravitz P, Cristea IA. Interpersonal Psychotherapy for Mental Health Problems: A Comprehensive Meta-Analysis. Am J Psychiatry. 2016 Jul 1;173(7):680-7. doi: 10.1176/appi.ajp.2015.15091141. Epub 2016 Apr 1. PMID 27032627
- [Background] Ravitz P, Watson P, Lawson A, Constantino MJ, Bernecker S, Park J, Swartz HA. Interpersonal Psychotherapy: A Scoping Review and Historical Perspective (1974-2017). Harv Rev Psychiatry. 2019 May/Jun;27(3):165-180. doi: 10.1097/HRP.0000000000000219. PMID 30883446
- [Background] Pu J, Zhou X, Liu L, Zhang Y, Yang L, Yuan S, Zhang H, Han Y, Zou D, Xie P. Efficacy and acceptability of interpersonal psychotherapy for depression in adolescents: A meta-analysis of randomized controlled trials. Psychiatry Res. 2017 Jul;253:226-232. doi: 10.1016/j.psychres.2017.03.023. Epub 2017 Mar 16. PMID 28391140
- [Background] Poleshuck EL, Talbot NE, Zlotnick C, Gamble SA, Liu X, Tu X, Giles DE. Interpersonal psychotherapy for women with comorbid depression and chronic pain. J Nerv Ment Dis. 2010 Aug;198(8):597-600. doi: 10.1097/NMD.0b013e3181ea4d3d. PMID 20699727
- [Background] Palmer S, Vecchio M, Craig JC, Tonelli M, Johnson DW, Nicolucci A, Pellegrini F, Saglimbene V, Logroscino G, Fishbane S, Strippoli GF. Prevalence of depression in chronic kidney disease: systematic review and meta-analysis of observational studies. Kidney Int. 2013 Jul;84(1):179-91. doi: 10.1038/ki.2013.77. Epub 2013 Mar 13. PMID 23486521
- [Background] Tian N, Chen N, Li PK. Depression in dialysis. Curr Opin Nephrol Hypertens. 2021 Nov 1;30(6):600-612. doi: 10.1097/MNH.0000000000000741. PMID 34456238
- [Background] Gerogianni G, Kouzoupis A, Grapsa E. A holistic approach to factors affecting depression in haemodialysis patients. Int Urol Nephrol. 2018 Aug;50(8):1467-1476. doi: 10.1007/s11255-018-1891-0. Epub 2018 May 19. PMID 29779116
- [Background] Frasure-Smith N, Koszycki D, Swenson JR, Baker B, van Zyl LT, Laliberte MA, Abramson BL, Lambert J, Gravel G, Lesperance F. Design and rationale for a randomized, controlled trial of interpersonal psychotherapy and citalopram for depression in coronary artery disease (CREATE). Psychosom Med. 2006 Jan-Feb;68(1):87-93. doi: 10.1097/01.psy.0000195833.68482.27. PMID 16449416
- [Background] Belay W, Kaba M, Labisso WL, Tigeneh W, Sahile Z, Zergaw A, Ejigu A, Baheretibeb Y, Gufue ZH, Haileselassie W. The effect of interpersonal psychotherapy on quality of life among breast cancer patients with common mental health disorder: a randomized control trial at Tikur Anbessa Specialized Hospital. Support Care Cancer. 2022 Jan;30(1):965-972. doi: 10.1007/s00520-021-06508-y. Epub 2021 Aug 25. PMID 34432169
- [Background] Yator O, Kagoya M, Khasakhala L, John-Stewart G, Kumar M. Task-sharing and piloting WHO group interpersonal psychotherapy (IPT-G) for adolescent mothers living with HIV in Nairobi primary health care centers: a process paper. AIDS Care. 2021 Jul;33(7):873-878. doi: 10.1080/09540121.2020.1801981. Epub 2020 Aug 11. PMID 32781831
- [Background] Hedayati SS, Bosworth HB, Kuchibhatla M, Kimmel PL, Szczech LA. The predictive value of self-report scales compared with physician diagnosis of depression in hemodialysis patients. Kidney Int. 2006 May;69(9):1662-8. doi: 10.1038/sj.ki.5000308. PMID 16598203
- [Background] Çınar, S. (2009). Hemodiyaliz hastalarında psikososyal uyum ve etkileyen faktörlerin belirlenmesi. Nefroloji Hemşireliği Dergisi, 6(1-2), 22-28.
- [Background] Davison SN. Personalized Approach and Precision Medicine in Supportive and End-of-Life Care for Patients With Advanced and End-Stage Kidney Disease. Semin Nephrol. 2018 Jul;38(4):336-345. doi: 10.1016/j.semnephrol.2018.05.004. PMID 30082054
- [Background] Schulman-Green D, Jaser S, Martin F, Alonzo A, Grey M, McCorkle R, Redeker NS, Reynolds N, Whittemore R. Processes of self-management in chronic illness. J Nurs Scholarsh. 2012 Jun;44(2):136-44. doi: 10.1111/j.1547-5069.2012.01444.x. Epub 2012 May 2. PMID 22551013
- [Background] Kacaroglu Vicdan A, Gulseven Karabacak B. Effect of Treatment Education Based on the Roy Adaptation Model on Adjustment of Hemodialysis Patients. Clin Nurse Spec. 2016 Jul-Aug;30(4):E1-E13. doi: 10.1097/NUR.0000000000000215. PMID 27309790
- [Background] Webster AC, Nagler EV, Morton RL, Masson P. Chronic Kidney Disease. Lancet. 2017 Mar 25;389(10075):1238-1252. doi: 10.1016/S0140-6736(16)32064-5. Epub 2016 Nov 23. PMID 27887750
- [Background] Romagnani P, Remuzzi G, Glassock R, Levin A, Jager KJ, Tonelli M, Massy Z, Wanner C, Anders HJ. Chronic kidney disease. Nat Rev Dis Primers. 2017 Nov 23;3:17088. doi: 10.1038/nrdp.2017.88. PMID 29168475
- [Background] Kalantar-Zadeh K, Jafar TH, Nitsch D, Neuen BL, Perkovic V. Chronic kidney disease. Lancet. 2021 Aug 28;398(10302):786-802. doi: 10.1016/S0140-6736(21)00519-5. Epub 2021 Jun 24. PMID 34175022